CLINICAL TRIAL: NCT03038932
Title: Integrated Extreme Trait Analysis to Understand the Etiology of Eczema Herpeticum (ADRN-06)
Brief Title: Etiology of Eczema Herpeticum (EH)
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Atopic Dermatitis Research Network (Other); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DAIT ADRN-06
Record Dates: First submitted 2017-01-25; First posted 2017-02-01 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Eczema Herpeticum
Keywords: whole genome sequencing (WGS)
MeSH Terms: conditions — Kaposi Varicelliform Eruption

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Skin Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Discovery Cohort: A minimum of 50 recurrent Atopic Dermatitis with a history of Eczema Herpeticum(ADEH+), 500 Atopic Dermatitis without a history of Eczema Herpeticum (ADEH-), and 237 Non-Atopic (NA) European American participants from the Atopic Dermatitis Research Network (ADRN) DNA Repository.
  The study will learn from this cohort:
  1. All Single Nucleotide Variants (SNVs) in ADEH+
  2. ADEH+ specific deleterious SNVs
  The study will determine the function of:
  4. ADEH+ risk variants
- Independent populations of participants: Two independent populations of participants:
  1. Children, aged 3-17 years and
  2. Adults 18-64 years of age.
  A minimum of 12 recurrent Atopic Dermatitis with a history of Eczema Herpeticum (ADEH+) with ≥3 Eczema Herpeticum (EH) episodes, 12 Atopic Dermatitis without a history of Eczema Herpeticum (ADEH-) and 12 Non-Atopic (NA) participants will be enrolled in each of the two populations.

SUMMARY:
Atopic dermatitis, also called eczema, is a disease with dry, scaly, itchy skin. Those with atopic dermatitis may have complications from skin infections such as eczema herpeticum after herpes simplex virus (HSV) infection. Symptoms of eczema herpeticum include fever and clusters of itchy blisters which crust over and form sores. Although exposure to HSV is widespread, most people clear the virus and only a subset of individuals with atopic dermatitis develop eczema herpeticum.

The purpose of this study is to determine why some individuals with atopic dermatitis are at higher risk for recurrent skin infections with HSV. The study team will compare how people with atopic dermatitis with a history of recurrent eczema herpeticum, people with atopic dermatitis without a history of eczema herpeticum, and people without atopic dermatitis respond to HSV.

DETAILED DESCRIPTION:
This study uses whole genome sequencing (WGS) technology to identify genetic variants that confer risk of recurrent atopic dermatitis with a history of eczema herpeticum (ADEH+), with ≥3 eczema herpeticum (EH) episodes.

A small subgroup of individuals with atopic dermatitis (AD) suffer from life-threatening disseminated herpes simplex virus (HSV) skin infections, termed eczema herpeticum (ADEH+). The manifestation of ADEH+ however is not simply a consequence of herpes simplex virus type 1 (HSV-1) infections, since the majority of the US population is latently infected with HSV-1 from an early age. Most importantly, there is a bimodality in the recurrence of eczema herpeticum (EH) episodes; most individuals have only a single episode but a subgroup of ADEH+ individuals has 3 or more episodes.

This study aims to conduct an extreme trait investigation of ADEH+ with recurrent EH, ≥3 episodes, compared to AD without a history of eczema herpeticum (ADEH-), using whole genome sequencing.

ELIGIBILITY:
Inclusion Criteria:

1. Must be a participant already enrolled in the ADRN Registry and provided DNA (ClinicalTrials.gov ID: NCT01494142);
2. Participant and/or parent guardian must be able to understand and provide informed consent;
3. A history of Atopic Dermatitis (AD) with a history of eczema herpeticum (ADEH+), as diagnosed using the Atopic Dermatitis Research Network (ADRN) Standard Diagnostic Criteria, with ≥3 episodes of Eczema Herpeticum (EH)

   OR

   A history of AD without a history of eczema herpeticum (ADEH-), as diagnosed using the ADRN Standard Diagnostic Criteria, and no immediate family members (mother, father, full siblings, half-siblings, offspring, aunts, uncles, cousins, or grandparents) with a history of EH

   OR

   Non-atopic as diagnosed using the ADRN Standard Diagnostic Criteria.
4. Anti-Herpes Simplex Virus (HSV)-1 or Anti-HSV-2 Immunoglobulin G (IgG) seropositive.

Exclusion Criteria:

1. Inability or unwillingness of a participant and/or parent guardian to give written informed consent or comply with study protocol;
2. Pregnant or lactating women;
3. Known or suspected immunosuppression;
4. Severe concomitant illness(es);
5. History of keloid formation (adults only);
6. History of lidocaine or Novocain allergy (adults only);
7. History of serious life-threatening reaction to latex, tape, or adhesives;
8. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.
9. Use of biologics within 5 half-lives (if known) or 16 weeks of the Screening Visit;
10. Use of an investigational drug within 5 half-lives (if known) or 8 weeks of the Screening Visit.

Ages: 3 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A minimum of 50 recurrent Atopic Dermatitis with a history of Eczema Herpeticum(ADEH+), 500 Atopic Dermatitis without a history of Eczema Herpeticum (ADEH-), and 237 Non-Atopic (NA) European American participants from the Atopic Dermatitis Research Network (ADRN) DNA Repository. The protocol will also enroll two independent populations of participants 1) children, 3-17 years of age and 2) adults 18-64 years of age. A minimum of 12 recurrent ADEH+ with ≥3 EH episodes, 12 ADEH- and 12 NA participants will be enrolled in each of the two populations.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
The Difference in Frequency of Rare Deleterious Coding Genetic Variants between Subjects with Recurrent Atopic Dermatitis (AD) and a History of Eczema Herpeticum (ADEH+) Compared to Controls - Using Whole Genome Sequencing | 3 years
  Whole genome sequencing methodology will be used to identify differences in frequency of rare deleterious coding genetic variants between recurrent Atopic Dermatitis (AD) subjects with a history of Eczema Herpeticum (ADEH+) and ≥3 Eczema Herpeticum (EH) episodes, versus controls. Controls will include (1) AD subjects without a history of EH (ADEH-); (2) non-atopic (NA) subjects without AD; and (3) general population controls from the Thousand Genomes Project.
The Difference in Frequency of Rare Deleterious Non-Coding Genetic Variants between Subjects with Recurrent Atopic Dermatitis (AD) and a History of Eczema Herpeticum (ADEH+) Compared to Controls - Using Whole Genome Sequencing | 3 years
  Whole genome sequencing methodology will be used to identify differences in frequency of rare deleterious non-coding genetic variants between subjects with recurrent Atopic Dermatitis (AD) subjects and a history of Eczema Herpeticum (ADEH+) with ≥3 Eczema Herpeticum (EH) episodes, versus controls. Controls will include (1) AD subjects without a history of EH (ADEH-); (2) non-atopic (NA) subjects without AD; and (3) general population controls from the Thousand Genomes Project.

SECONDARY OUTCOMES:
Gene expression profiles in the dermis | 3 years
Gene expression profiles in the epidermis | 3 years
Gene expression profiles in in keratinocytes | 3 years
Gene expression profiles in fibroblasts | 3 years
Gene expression profiles in peripheral blood Plasmacytoid Dendritic Cells(pDCs) | 3 years
Gene expression profiles in skin tape strip samples | 3 years
Herpes Simplex Virus (HSV) replication in primary keratinocytes | 3 years
  HSV replication will be assessed by HSV copy number by Polymerase Chain Reaction (PCR) or RNA sequencing.
Herpes Simplex Virus (HSV) replication in fibroblasts | 3 years
  HSV replication will be assessed by HSV copy number by Polymerase Chain Reaction (PCR) or RNA sequencing.
Herpes Simplex Virus (HSV) replication in Plasmacytoid Dendritic Cells (pDCs) | 3 years
  HSV replication will be assessed by HSV copy number by Polymerase Chain Reaction (PCR) or RNA sequencing.
Herpes Simplex Virus (HSV) replication in genetically modified cell lines | 3 years
  HSV replication will be assessed by HSV copy number by Polymerase Chain Reaction (PCR) or RNA sequencing.
Anti-viral responses in primary keratinocytes | 3 years
  Anti-viral responses will be measured by cytokine production and antimicrobial responses (e.g. interferons [IFNs], tumor necrosis factor alpha [TNFalpha], LL-37, human beta-defensins [HBDs])
Anti-viral responses in fibroblasts | 3 years
  Anti-viral responses will be measured by cytokine production and antimicrobial responses (e.g. interferons [IFNs], tumor necrosis factor alpha [TNFalpha], LL-37, human beta-defensins [HBDs])
Anti-viral responses in Plasmacytoid Dendritic Cells (pDCs) | 3 years
  Anti-viral responses will be measured by cytokine production and antimicrobial responses (e.g. interferons [IFNs], tumor necrosis factor alpha [TNFalpha], LL-37, human beta-defensins [HBDs]).
Anti-viral responses in genetically modified cell lines | 3 years
  Anti-viral responses will be measured by cytokine production and antimicrobial responses (e.g. interferons [IFNs], tumor necrosis factor alpha [TNFalpha], LL-37, human beta-defensins [HBDs]).
Immune responses in primary keratinocytes | 3 years
  Immune responses will be measured by cytokine production and antimicrobial responses (e.g. interferons [IFNs], tumor necrosis factor alpha [TNFalpha], LL-37, human beta-defensins [HBDs]).
Immune responses in fibroblasts | 3 years
  Immune responses will be measured by cytokine production and antimicrobial responses (e.g. interferons [IFNs], tumor necrosis factor alpha [TNFalpha], LL-37, human beta-defensins [HBDs]).
Immune responses in Plasmacytoid Dendritic Cells (pDCs) | 3 years
  Immune responses will be measured by cytokine production and antimicrobial responses (e.g. interferons [IFNs], tumor necrosis factor alpha [TNFalpha], LL-37, human beta-defensins [HBDs]).
Immune responses in genetically modified cell lines | 3 years
  Immune responses will be measured by cytokine production and antimicrobial responses (e.g. interferons [IFNs], tumor necrosis factor alpha [TNFalpha], LL-37, human beta-defensins [HBDs])
Differentiation markers in primary keratinocytes | 3 years
  Differentiation markers (e.g. filaggrin (FLG), involucrin, loricrin, and Human Beta-Defensins (HBDs)).
Differentiation markers in genetically modified keratinocyte cell lines | 3 years
  Differentiation markers (e.g. filaggrin (FLG), involucrin, loricrin, and Human Beta-Defensins (HBDs)).
Expression of reporter gene constructs testing non-coding variants | 3 years
Exploratory: Viral carriage | 3 years
  Viral carriage will be assessed by presence of viral sequencing reads.
Exploratory: Protein expression of epidermal differentiation complex | 3 years
  Protein expression of epidermal differentiation complex will be measured by Mass Spectroscopy of skin tape strips.
Exploratory: Protein expression of inflammatory genes | 3 years
  Protein expression of inflammatory genes will be measured by Mass Spectroscopy of skin tape strips.
Exploratory: Lipid profiles | 3 years
  Lipid profiles will be measured by mass spectroscopy of skin tape strips.
Exploratory: Whole-genome DNA methylation profiles from epidermis | 3 years
Exploratory: Whole-genome DNA methylation profiles from dermis | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Donald Leung, M.D., Ph.D., Study Chair — National Jewish Health: Division of Pediatric Allergy and Clinical Immunology
Locations (1):
- National Jewish Health: Division of Pediatric Allergy and Clinical Immunology, Denver, Colorado, United States

REFERENCES:
- See also: ClinicalTrials.gov Record for Atopic Dermatitis Research Network Registry — https://clinicaltrials.gov/ct2/show/NCT01494142
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Atopic Dermatitis Research Network (ADRN) information — https://www.niaid.nih.gov/research/atopic-dermatitis-research-network